CLINICAL TRIAL: NCT04848246
Title: Efficacy of Smoking Cessation Interventions on Tuberculosis Treatment Outcomes Among Newly Diagnosed Pulmonary Tuberculosis Patients; a Single Blind Randomized Controlled Trial
Brief Title: Effect of Smoking Cessation on Tuberculosis Treatment Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Muhammad Tahir Rizwan Khan, Assistant Professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-898/DUHS/Approval/2017/136
Record Dates: First submitted 2021-04-04; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Tuberculosis, Pulmonary
Keywords: smoking cessation
MeSH Terms: conditions — Tuberculosis, Pulmonary; Smoking Cessation | interventions — Bupropion

STUDY DESIGN:
Intervention Model Description: A total of three groups, two intervention and one control
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor for tuberculosis outcomes at the study site were blinded in terms of intervention allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bupropion (Experimental)
  Interventions: Drug: Bupropion; Behavioral: Behavioural Change Communication
- Behavioural Change Communication (Experimental)
  Interventions: Behavioral: Behavioural Change Communication
- Control (No Intervention)

INTERVENTIONS:
Drug: Bupropion — This group received Bupropion 150 mg twice daily for 10 weeks
  Arms: Bupropion
Behavioral: Behavioural Change Communication — This group will receive Behavioural Change Communication
  Arms: Behavioural Change Communication; Bupropion

SUMMARY:
This study was a Randomized Controlled Trial conducted at Ojha Institute of Chest Diseases, Dow University of Health Sciences, Karachi, among pulmonary tuberculosis patients

ELIGIBILITY:
Inclusion Criteria:

* pulmonary tuberculosis patients of age 18 years or above
* registered under Directly Observed Treatment Short course (DOTS) at Ojha Institute of Chest Diseases
* reported to have smoked 100 plus cigarettes in past and currently smoking cigarettes

Exclusion Criteria:

* Extra pulmonary tuberculosis
* drug resistant tuberculosis
* pregnancy
* positive history of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Percentage of patients completing anti-tuberculosis treatment | six months
  Among both smear positive and smear negative TB patients, successful completion of ATT will be labeled at the end of 6 months period if the patients has been compliant with ATT through six months period..

SECONDARY OUTCOMES:
Percentage of participants achieving abstinence from smoking | six months
  Abstinence is defined as staying away from smoking and it will be assessed at week 1, week 4, week 12 and week 24 will be assessed in following two ways:
  i. Self-reported abstinence using questionnaire ii. Expired carbon monoxide (eCO) levels using Micro Smokerlyzer (Bedfont Scientific) of less than 7 ppm.

OTHER OUTCOMES:
Percentage of patients defaulting anti-tuberculosis treatment. | Six Months
  Treatment default will be defined as interruption of anti-tuberculosis treatment for ≥2 consecutive months. This outcome will be assessed in both smear positive and smear negative patients.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Tahir Rizwan Khan, M.Phil., Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No